CLINICAL TRIAL: NCT03305861
Title: GreenLight (532nm) LASER (XPS) Enucleation vs. Thulium LASER Enucleation of Prostate for Treatment of Benign Prostatic Hyperplasia
Brief Title: Green LEP vs ThuLEP in Management of Marked Enlarged Prostate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Laymon, MD, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD/17.02.26
Record Dates: First submitted 2017-09-22; First posted 2017-10-10 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Prostatic Hyperplasia With Urinary Obstruction
Keywords: Thulium Laser Enucleation of the Prostate (ThuLEP); Greenlight Laser Enucleation of the Prostate (Green LEP)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ThuLEP (Experimental): Thulium laser enucleation of prostate
  Interventions: Procedure: ThuLEP
- Green LEP (Experimental): Greenlight laser enucleation of prostate
  Interventions: Procedure: Green LEP

INTERVENTIONS:
Procedure: ThuLEP — Thulium laser enucleation of prostate
  Arms: ThuLEP
Procedure: Green LEP — Greenlight laser enucleation of prostate
  Arms: Green LEP

SUMMARY:
In this study the investigators aim to test TGreenlight (532-nm) laser Photoselective Enucleation of the Prostate (Green LEP) using (XPS) 180W system ) vs Thulium Laser 200 W Enucleation of the Prostate (ThuLEP) in reduction of lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH) in a randomized controlled trial. Furthermore, all peri-operative parameters, urinary flow parameters, prostate size changes and complications associated with the procedures will be compared.

DETAILED DESCRIPTION:
Transurethral resection of the prostate (TURP) and open simple prostatectomy (SP) have been the historical reference-standard procedures for prostates < 80 g and ≥ 80 to 100 g, respectively, for years.

Evolution of LASER technology revived the concept of enucleation, so that the resectoscope can be used instead of the surgeon's index finger to separate the adenoma from the surgical capsule mimicking OP. There are several types of laser energy available for enucleation, but the commonest types are Holmium, Greenlight (532nm) and Thulim YAG LASERS.

Thulium: yttrium-aluminium-garnet laser Thulium LASER works at a wavelength between 1940 and 2013 nm in continuous wave mode so it offers advanced vaporization and hemostatic features. Different applications and techniques were developed ranging from vapoenucleation technique with in situ laser assisted resection, so-called Tangerine technique (Thulium Laser resection of the prostate Tangerine Technique "TmLRP-TT"), and enucleation (ThuVEP/ThuLEP are published.

Inspite of paucity of RCT comparing ThuLEP to other standard techniques in management of large prostate, long term outcomes of ThuLEP are so robust. Gross et al reported their 5 year follow up after ThuVEP in 500 patients with median prostate size of 50 grams. They demonstrated durable outcomes, with persistent reductions in I-PSS score (5 vs 21), QoL score (1 vs 4) and improvement in Q max (16.3 vs 6.9 ml/sec). Late complications included urethral stricture in 3.1%, BNC in 3.1% and recurrent adenoma in 0.6%.

Yang et al published their 5 year results of a RCT comparing ThuLEP vs TURis in 159 patients with median prostate size of 70 gm. No statistically significant difference between both groups in terms of IPSS, Qmax or post voiding residual. No patient in either group required retreatment.

In RCT by Feng et al comparing ThuLEP to PKEP ,with 18 months follow up results , the former proved to be efficient and safe within 12 months follow-up interval. However, ThuLEP had significantly better hemostasis parameters and shorter catheterization time.

III GreenLight (532nm) laser system

The Kalium-Titanyl-Phosphate (KTP) and the lithium triborate (LBO) lasers work at a wavelength of 532 nm. Laser energy is absorbed by haemoglobin, but not by water. Vaporisation leads to immediate removal of prostatic tissue, relief of BPO, and reduction of LUTS. GreenLight laser has gained increasing acceptance as a less invasive treatment for lower urinary tract symptoms due to benign prostatic hyperplasia (BPH/ LUTS).

A meta-analysis of the nine available RCTs comparing PVP using the 80-W and 120-W lasers with TURP , no differences were found in Qmax and IPSS between 80-W-PVP and TURP, but only two RCTs provided sufficient 12-month data to be included in the meta-analysis.

With the 180-W (XPS) laser efficacy is comparable to TURP in terms of IPSS, Qmax, post voided residual volume, prostate volume reduction, PSA decrease and QoL questionnaires. The XPS laser prostatectomy is superior to TURP in terms of catheterisation time, lengths of hospital stay and time to stable health status.

In a RCT by Al-Ansari et al comparing HPS 120-W laser PVP versus TURP , the former was associated with dramatic improvements in all urinary outcomes compared to TURP, but reintervention rate for recurrent adenomas was 11 % compared to 1.8% in TURP group. All patients who needed redo surgery had prostate larger than 80 gm.

In another RCT, El-Shal et al of a compared Greenlight laser 180W XPS vapo enucleation , where the adenoma is bluntly enucleated partially then vaporized in situ, and HoLEP and reported 12 months follow up results. Green light XPS vapoenucleation was comparable and non inferior to HoLEP in symptom improvement. However, at 12 months Q max, prostate size reduction and PSA reduction were significantly higher in HoLEP group.

These important findings highlighted some limitations in PVP or vapoenucleation such as the difficulty in determining the anatomical cleavage limits and capsular plain of large adenomas. These drawbacks are not related to the energy source but to the technique used.

Gomez Sancha described different technique to avoid these limitations which was Greenlight LASER En-bloc Enucleation of Prostate (Green LEP) where the whole adenoma is dissected from the surgical capsule and morcellated at the end.

Misrai et al compared Green LEP vs Greenlight PVP for management of prostates larger than 80 gms. At 6 months follow up, IPSS, QoL and PVR improved similarly in both groups but Q max was significantly higher in Green LEP group. Median percent reduction in prostate size as measured by TRUS was significantly higher in green LEP (74% vs 57%). Median % reduction of PSA was 40% and 67% in PVP and Green LEP respectively (p<0.0001).

There is a paucity in studies comparing different types of EEP using different energy sources other than holmium laser.

Aim of the work In this study the investigators aim to test Thulium Laser 200 W Enucleation of the Prostate (ThuLEP) vs Greenlight (532-nm) laser Photoselective Enucleation of the Prostate (Green LEP) using (XPS) 180W system in reduction of LUTS secondary to BPH in a randomized controlled trial. Furthermore, all peri-operative parameters, urinary flow parameters, prostate size changes and complications associated with the procedures will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ≥ 40 years
* LUTS secondary to BOO due to BPH who failed medical treatment
* International prostate symptom scores (IPSS) >15 and bother score (QOL) ≥ 3 (according to IPSS question 8)
* Peak urinary flow rate (Qmax) <15 ml/sec with at least 125 ml voided volume or Patients with acute urine retention secondary to BPH who failed trial of voiding on medical treatment.
* ASA (American society of anaesthesiologists) score ≤3.
* TRUS prostate size > /= 80 ml

Exclusion Criteria:

* Patient with neurological disorder which might affect bladder function as cerebrovascular stroke, Parkinson disease
* Active urinary tract infection,
* Presence of active bladder cancer (within the last 2 years)
* Known prostate cancer patients will be excluded preoperatively on the basis of digital rectal examination, prostate specific antigen level, and TRUS imaging followed by prostate biopsies if necessary.
* Patient has a disorder of the coagulation cascade (e.g., liver cell failure) or disorders that affect platelet count or function (e.g., von Willebrand disease) that would put the subject at risk for intraoperative or postoperative bleeding.
* Patient is unable to discontinue anticoagulant and antiplatelet therapy preoperatively (3-5 d) except for low-dose aspirin (e.g., 100 mg).
* Patient has had an acute myocardial infarction or open-heart surgery <180 days prior to the date of informed consent.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
voiding and storage symptoms improvement | 6 months
  International Prostate Symptom Score (I-PSS)
sexual function changes | 6 months
  International Index of Erectile Function Questionnaire (IIEF)

SECONDARY OUTCOMES:
Operative time | 6 months
  in minutes
Postoperative complication | 12 months
  Clavien-Dindo classification for post-operative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Dakahlia Governorate, Egypt